CLINICAL TRIAL: NCT02256358
Title: Comparison of Effects of Intravenous Midazolam and Ketamine on Emergence Agitation : a Randomized Controlled Trial
Brief Title: Comparison of Effects of Intravenous Midazolam and Ketamine on Emergence Agitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Ki Hwa Lee, Assistant professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2012-127
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Psychomotor Agitation
Keywords: child, ketamine, midazolam
MeSH Terms: conditions — Psychomotor Agitation | interventions — Midazolam; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam (Active Comparator): Intravenous 0.1 mg/kg midazolam was administered to the patients as premedication drug before entering operating room.
  Interventions: Drug: Midazolam
- Ketamine (Experimental): Intravenous 1 mg/kg ketamine was administered to the patients as premedication drug before entering operating room.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Midazolam — preoperatively injected intravenous 0.1 mg/kg midazolam
  Arms: Midazolam
Drug: Ketamine — Preoperatively injected intravenous 1mg/kg ketamine
  Other Names: Ketamine HCl
  Arms: Ketamine

SUMMARY:
Compare the effects of intravenous midazolam and ketamine on emergence agitation after sevoflurane anesthesia

DETAILED DESCRIPTION:
Emergence agitation is self-limiting aggressive behavior that develops in the early period of awakening from anesthesia. A high level of preoperative anxiety is a risk factor for emergence agitation using Aono's four-point scale. Midazolam and ketamine was administered to the patients to decrease of preoperative anxiety. We aimed to compare the emergence agitation between midazolam group and ketamine group.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists physical status 1-2 aged 2-6 years old, who were scheduled to undergo ophthalmic surgery (<2hr)

Exclusion Criteria:

* children with central nervous system disorders,history of allergy to the study drugs (midazolam and ketamine), history of recent respiratory tract infection

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kihwa Lee, MD, Study Chair — Haeundae paik hospital, inje university

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Midazolam | Ketamine
Started | 34 | 34
Completed | 34 | 33
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam | Ketamine | Total
Number analyzed (Participants) | 34 | 33 | 67
Age, Continuous [Mean (Standard Deviation); unit: year] | 4.15 (1.40) | 4.21 (1.32) | 4.18 (1.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Emergence Agitation
Description: The primary endpoint is the incidence of postoperative emergence agitation that was defined as an Aono's four-point scale(AFPS) score of 3 or higher.
Time Frame: During 30 minutes after extubation at post-anesthetic care unit, every 5 minutes
Measure: Number; unit: participants
Arm/Group | Midazolam | Ketamine
Number analyzed (Participants) | 34 | 33
participants | 6 | 0

ADVERSE EVENTS:
Time Frame: 1 day
Description: Recording of complications at 5 minutes intervals during 30 minutes after operation
Arm/Group | Midazolam | Ketamine
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 0/34 | 0/34

LIMITATIONS AND CAVEATS:
We did not include a placebo group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No